CLINICAL TRIAL: NCT00731887
Title: Assessment of the Treatment of the Severely Burned With Anabolic Agents on Improved Wound Healing, Recovery and Rehabilitation: Large Burn Outcome Study
Brief Title: Large Burn Outcome Study
Acronym: LBO
Status: Withdrawn | Type: Observational
Why Stopped: Personnel involved in this protocol are no longer associated with this study
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Other Study IDs: 04-157B
Record Dates: First submitted 2008-07-30; First posted 2008-08-11 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-12

CONDITIONS: Burns
Keywords: Burn injury; Burn recovery
MeSH Terms: conditions — Burns | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine collected for this study will be retained for possible re-analysis if needed for the duration of the study.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood and urine testing — complete blood count, routine chemistries, liver function test, retinol binding protein, transferrin, prothrombin time, partial thromboplastin time, fibrinogen, Vitamin A and Zinc, Insulin Growth Factor levels and binding proteins, cytokines (interleukins 1, 6, 12), insulin, thyroid hormones, cortisol, 25-hydroxyvitamin D, and osteocalcin.

SUMMARY:
To examine long term physical and psychosocial outcomes of pediatric burn survivors. We want to learn about thoughts, feelings, coping style, social support, and overall adjustment following burn injury.

DETAILED DESCRIPTION:
To evaluate the long term quality of life of adolescents and adults who suffered severe pediatric burns. This study will include an array of physical and psychosocial assessments, thus providing a unique and complete set of information on the long term outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* At least 60% third degree total body surface area
* Acute burn treatment at Shriners Burns Hospital for Children - Galveston between 1986-2005
* Three years post injury
* Current age of at least 16 years

Exclusion Criteria:

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those that have received a burn injury at least 3 years ago and that recieved acute burn treatment at Shriners Hospital for Children - Galveston between 1986-2005.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas